CLINICAL TRIAL: NCT00992693
Title: Treatment of Viral Hemorrhagic Fever (Crimean-Congo Hemorrhagic Fever or Lassa Fever) With Intravenous Ribavirin in Department of Defense (DOD) Associated Medical Treatment Facilities: A Phase 2 Study
Brief Title: Treatment of Viral Hemorrhagic Fevers With Intravenous Ribavirin in Military Treatment Facilities
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C2009.140
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-09

CONDITIONS: Crimean-Congo Hemorrhagic Fever; Lassa Fever
Keywords: Crimean-Congo Hemorrhagic Fever; Lassa Fever; CCHF; LF; Viral Hemorrhagic Fever; VHF; Ribavirin
MeSH Terms: conditions — Hemorrhagic Fever, Crimean; Lassa Fever; Hemorrhagic Fevers, Viral | interventions — Ribavirin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with IV Ribavirin (Experimental): In this open label treatment study, the investigators intend to treat all subjects who present with a tentative diagnosis of VHF and meet entry criteria with a 10 day course of IV Ribavirin.
  Interventions: Drug: Ribavirin (Virazole) Injection

INTERVENTIONS:
Drug: Ribavirin (Virazole) Injection — The drug is to be administered in a volume of 50-100 ml of normal saline to be infused over 30-40 minutes.
  1) Loading dose: 33 mg/kg (maximum dose 2.64 g)(1 dose) 2) Followed by a dose of 16 mg/kg (max dose 1.28 g) every 6 hours for the first 4 days (15 doses) 3) Followed by a dose of 8 mg/kg (maximum dose 0.64 g) every 8 hours for the subsequent 6 days (18 doses) Ten day course of treatment with follow up between day 28 to day 60.
  Other Names: Virazole Injection, 100 mg/ml

SUMMARY:
This is a Phase 2 study of the safety and efficacy of Intravenous (IV) Ribavirin in treating patients presenting with a probable or suspected case of viral hemorrhagic fever (either Crimean Congo or Lassa Fever) at a military medical treatment hospital. All patients will be treated with a 10 day course of IV Ribavirin if they meet all the inclusion and none of the exclusion criteria.

DETAILED DESCRIPTION:
Department of Defense operations have resulted in the deployment of personnel to areas endemic for Viral Hemorrhagic Fever (VHF): Crimean-Congo Hemorrhagic Fever (CCHF) or Lassa Fever. Unfortunately, beyond supportive care, there is no approved therapy for treating either infection. Previous studies with intravenous (IV) Ribavirin have shown IV Ribavirin as a promising treatment for both infections. This study will provide experience in U.S. Department of Defense associated treatment facilities in the use of IV Ribavirin for the experimental treatment of viral hemorrhagic fevers primarily among U.S. Service personnel deployed to disease-endemic areas.

The rationale for conducting the study is a) to allow the DoD to gain experience in treating VHF b) to offer this experimental but promising therapy to patients with probable or suspected VHF c) to collect safety data while obtaining experience using Ribavirin.

ELIGIBILITY:
Inclusion Criteria:

An individual will be enrolled in this study if the patient:

* Meets the case definition for a probable or a suspected case of CCHF or LF (see below).
* Has read and signed the Informed Consent.
* Is at least 18 years of age (17, if active military) and not greater than 65 years of age.
* Has a blood sample drawn and a type and cross-match ordered for transfusion.
* Agrees to collection of required specimens.
* Agrees to report any Adverse Events, Serious and Unexpected Adverse Events for the duration of the study.
* Agrees to a follow-up visit and to donate blood and urine specimens at day 14 (±2 days) and once between days 28 and 60 after the first dose of IV Ribavirin and to all follow-up visits for anemia or other medical conditions as required by the attending physician.
* Woman of childbearing age must have a pregnancy test performed. If negative, she must agree not to become pregnant during treatment and for 7 months after receiving Ribavirin. She also must agree to not breast feed during treatment and for 7 months after receiving Ribavirin. Two reliable forms of effective contraception must be used including one barrier method during treatment and during the 7 month post-treatment period. She will be counseled concerning the risks of IV Ribavirin versus no treatment if the pregnancy test is positive.
* Man agrees not to have intercourse with pregnant woman during treatment and for 7 months after receiving Ribavirin, and take precautions to avoid producing pregnancies during treatment and for 7 months after receiving Ribavirin. At least two reliable forms of effective contraception must be used including one barrier method during treatment and during the 7 month post-treatment period to avoid a pregnancy.
* Has a hemoglobin greater than or equal to10 g/dL before starting IV Ribavirin

Note: Malaria should be excluded as a possibility for illness in patients suspected to have VHF.

Probable Case of Crimean-Congo Hemorrhagic Fever:

All subjects will have a history of possible exposure to CCHF, either having:

* Worked or slept outdoors in the CCHF endemic area within 2 weeks of illness onset, with or without a history of tick-bite or tick exposure, (Endemic area includes, but not necessarily limited to: Saudi Arabia, Kuwait, Oman, United Arab Emirates, Iran, Iraq, Turkey, Greece, Bulgaria, Albania, Montenegro, the Kosovo region of Serbia, Bosnia-Herzegovina, Macedonia, the whole of Africa, India, Pakistan, Afghanistan, Kazakhstan, Uzbekistan, Kyrgyzstan, Tajikistan, Turkmenistan, Azerbaijan, Georgia, the Crimean region of the Ukraine, Rostov-Don and Astrakhan regions of Russia, and the Xinjiang [northwestern] region of the People's Republic of China), OR
* Handled blood or freshly butchered meat of domestic livestock in CCHF endemic area during 2 weeks before the onset of illness, OR
* Had direct contact with blood, tissues, secretions, or excretions of a CCHF patient (suspected or confirmed), including laboratory specimens, OR
* Worked with the virus in the laboratory setting and have a clinical syndrome consistent with CCHF as defined by:

  * Acute illness with fever and at least two of these symptoms: myalgia, low back pain, and headache,
  * And the appearance of three or more of the following five groups of signs/symptoms:

    * Hemorrhage (one or more petechiae, ecchymoses, purpura, gingival bleeding, epistaxis, gastrointestinal tract bleeding),
    * Elevated AST levels (above the upper limits of normal for the laboratory),
    * Thrombocytopenia (below the lower limits of normal),
    * Hypotension (systolic pressure < 90 mm Hg), or
    * Azotemia, renal failure (serum creatinine above the upper limits of normal).
* Prognostic indicators exist for subjects at increased risk of severe CCHF. Any of these indicators occurring in the first 5 days of illness, predict a mortality greater than 90% (Swanepoel et al., 1989). Patients with these prognostic indicators may benefit most from drug therapy, if resources become limiting:

  * WBC > 10,000/mm3
  * Platelet count < 20 x 103/mm3
  * AST > 200 U/L
  * ALT > 150 U/L
  * APTT > 60 seconds
  * Fibrinogen < 110 mg/dL

Probable Case of Lassa Fever:

All subjects will have a history of possible exposure to Lassa fever, either having:

* By residence or travel in an endemic area where contact with rodents was possible within 3 weeks of onset of illness, (Endemic area includes, but not necessarily limited to: Sierra Leone, Liberia, Nigeria, Mali, Central African Republic, and Guinea.) or
* Contact with a suspect patient or their body fluids (including laboratory specimens) within 3 weeks of symptom onset, or
* Worked with the virus in the laboratory setting. And have
* A negative malaria smear. And have
* Signs and symptoms compatible with Lassa fever, either:

  * Fever plus pharyngitis plus retrosternal pain plus proteinuria (positive predictive value of 81% when these three criteria are met, McCormick et al., 1987a,b),OR
  * Fever plus unexplained mucosal bleeding, OR
  * Fever plus unexplained edema of the face and neck, OR
  * Suspected Case of CCHF or LF
* Have a clinical syndrome consistent with CCHF or LF, meeting most of the above criteria of a probable case and the patient has an epidemiological history of potential exposure to the bunyavirus or arenavirus (i.e., recent field duty and/or other individuals in his troop have CCHF or LF).

Exclusion Criteria:

* Has known intolerance to Ribavirin.
* Is irreversibly ill on presentation, as defined by presence of profound shock (shock which does not respond to supportive therapy within 3 hours after admission).
* Has hemoglobin less than 10 g/dL that cannot be corrected to 10 g/dL before initiation of IV Ribavirin
* Has history of hemoglobinopathies (i.e., sickle-cell anemia or thalassemia major).
* Has history of autoimmune hepatitis.
* Has a calculated serum creatinine clearance of < 30 mL/min.
* History of such as second or third degree heart block or sick sinus syndrome and without a pacemaker and no capability of a pacemaker placement or Wolfe-Parkinson-White Syndrome.
* A sinus bradycardia of less than 40 beats per minute.
* Is currently being treated with Didanosine (ddI). ddI must be discontinued before starting IV Ribavirin.

Relative Exclusion Criteria:

At the principal investigator's (PI) discretion, an individual may be treated with IV Ribavirin, with caution, if one of these criteria is present:

* A positive pregnancy test. The individual will be informed of the risk and benefit of treatment with IV Ribavirin versus no treatment with IV Ribavirin in CCHF (generally associated with high mortality) and severe cases of Lassa fever with high mortality rates versus mild cases of Lassa fever with low mortality rates.
* A New York Heart Association Cardiac functional capacity of Class II or greater for ASHD and CHF.
* Known cardiac defects that my predispose the subject to bradyarrhythmias, such as second or third degree heart block or sick sinus syndrome without a pacemaker, but capability of pacemaker placement, if needed.
* Sinus bradycardia of 41-49 beats per minutes if the individual is not known to have a low resting heart rate related to physical conditioning.
* Use of drugs known to result in bradyarrhythmias (certain betablockers and calcium channel blockers, digoxin).

  f. History of gout or tophaceous gout.

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2016-07-19 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 5 years
Number of deaths of individuals with viral hemorrhagic fever (Crimean-Congo hemorrhagic fever or Lassa fever) who received at least four doses of IV Ribavirin | 5 years

SECONDARY OUTCOMES:
Number of clinical events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Rini, MD, Principal Investigator — Landstuhl Regional Medical Center, Germany
Locations (1):
- Landstuhl Regional Medical Center, Landstuhl, Rhineland-Palatinate, Germany